CLINICAL TRIAL: NCT04495335
Title: The Effect of Photobiomodulation Application on Implant Stabilization and Peri-implant Microbiology
Brief Title: Photobiomodulation and Implant Stability
Acronym: low-laser
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: T.C. Dumlupınar Üniversitesi (Other)
Collaborators: Gazi University (Other)
Responsible Party: Principal Investigator, Berceste Guler, DDS PhD, Assist Prof, T.C. Dumlupınar Üniversitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-04/01
Record Dates: First submitted 2020-07-26; First posted 2020-07-31 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Photobiomodulation Therapy
Keywords: Low-level laser therapy implants
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Implants were randomly divided into two groups and implants placed in the test group were treated with Gallium-aluminum-arsenate (GaA1As) diode laser with photobiomodulation therapy immediately after surgery and for 15 days. In the control group, implants were not irradiated.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (TG) (Experimental): The study included test group with Photobiomodulation treatment after dental implant surgery
  Interventions: Device: photobiomodulation
- Control Group (CG) (Active Comparator): The control group consisted of laser application without energy delivery to the tissue.
  Interventions: Device: photobiomodulation

INTERVENTIONS:
Device: photobiomodulation — Laser treatment will complete using Gallium-Aluminum-Arsenide (GaA1As) diode laser and application will complete by laser energy immediately and three times a week for just 15 days after surgery.
  Other Names: low-level laser therapy

SUMMARY:
Objective: The aim of the present study was to address the following questions: does photobiomodulation therapy (PBMT) improve implant stability and affect microbiota around dental implants in the early stage of osseointegration.

Material and Methods: Implants will randomly be divided into two groups and implants will be placed in the test group treating with Gallium-aluminum-arsenate (GaA1As) diode laser with photobiomodulation therapy immediately after surgery and for 15 days. In the control group, implants are not irradiated. The primary stability of the implants will measure by the Resonance frequency analysis (RFA) after insertion and the secondary stability values will record at 30th, 60th, and 90th days after surgery as implant stability quotient (ISQ). Plaque samples will collect for microbiological analyzes at the first 24 hours after implant surgery and six days after 90 days at six sterile endodontic paper points.

DETAILED DESCRIPTION:
The same surgical procedure will be operated in the test and control groups by the same surgeon. Full-thickness flaps were raised and dental implant osteotomy preparation will be completed according to the manufacturers' instructions. Laser treatment will be completed using Gallium-Aluminum-Arsenide diode laser. The photobiomodulation application will v-be completed by laser energy immediately and three times a week for just 15 days after surgery. The control group will consist of laser application without energy delivery to the tissue. Immediately after implant placement, the third generation stability resonance frequency (RF) analyzer will be applied for direct measurement of implant stability and the value will be recorded. The microbiological plaque samples will be collected at specific times, according to the following schedule; at the first 24-hour and 90 days after implant surgery. All bacterial DNA specimen will be analyzed with qPCR technique to evaluate Aggregatibacter actinomycetemcomitans (Aa), Porphyromonas gingivalis (Pg), Prevotella intermedia (Pi) , Tannerella forsythia (Tf ) and total amount of bacteria.

ELIGIBILITY:
Inclusion Criteria:

* at least one tooth loss in left and right posterior sides of upper and lower jaws
* adequate alveolar bone volume as horizontal and vertical

Exclusion Criteria:

* uncontrolled systemic diseases
* parafunctional (bruxism and/or clenching)
* smoking habits
* any allergies or metabolic bone diseases,
* pregnancy
* surgical periodontal treatment in 6 months
* using antibiotics in the last 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
primary and secondary implant stability | The stability was measured at immediately postoperatively.
  Immediately after implant placement, the third generation stability resonance frequency (RF) analyzer (Osstell ISQ, Integration Diagnostics AB, Gamlestadsvägen, Goteborg, Sweden) was applied for direct measurement of implant stability and the value was recorded.
primary and secondary implant stability | The stability was measured at 30 days postoperatively.
  Immediately after implant placement, the third generation stability resonance frequency (RF) analyzer (Osstell ISQ, Integration Diagnostics AB, Gamlestadsvägen, Goteborg, Sweden) was applied for direct measurement of implant stability and the value was recorded.
primary and secondary implant stability | The stability was measured at 60 days postoperatively.
  Immediately after implant placement, the third generation stability resonance frequency (RF) analyzer (Osstell ISQ, Integration Diagnostics AB, Gamlestadsvägen, Goteborg, Sweden) was applied for direct measurement of implant stability and the value was recorded.
primary and secondary implant stability | The stability was measured at 90 days postoperatively.
  Immediately after implant placement, the third generation stability resonance frequency (RF) analyzer (Osstell ISQ, Integration Diagnostics AB, Gamlestadsvägen, Goteborg, Sweden) was applied for direct measurement of implant stability and the value was recorded.

SECONDARY OUTCOMES:
Evaluation of the number of peri-implant total microorganisms by PCR | Microbiological samples will obtained at the first 24-hour after implant surgery
  The sample of the dental implant to be sampled is gently isolated with sterile cotton rolls. Then standardized sterile endodontic paper-points with tip size 40 were inserted into crevice very gently avoiding gingival bleeding. The paper-points were immediately put into sterilized Eppendorf tubes.
Evaluation of the number of peri-implant total microorganisms by PCR | Microbiological samples will obtained at the 90 days after implant surgery
  The sample of the dental implant to be sampled is gently isolated with sterile cotton rolls. Then standardized sterile endodontic paper-points with tip size 40 were inserted into crevice very gently avoiding gingival bleeding. The paper-points were immediately put into sterilized Eppendorf tubes.

CONTACTS AND LOCATIONS:
Overall Officials: Suleyman Bozkaya, DDS PhD, Study Director — Gazi University Faculty of Dentistry
Locations (1):
- Kütahya Health Sciences University Faculty of Dentistry, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lioubavina-Hack N, Lang NP, Karring T. Significance of primary stability for osseointegration of dental implants. Clin Oral Implants Res. 2006 Jun;17(3):244-50. doi: 10.1111/j.1600-0501.2005.01201.x. PMID 16672018
- [Background] Kim YD, Kim SS, Hwang DS, Kim SG, Kwon YH, Shin SH, Kim UK, Kim JR, Chung IK. Effect of low-level laser treatment after installation of dental titanium implant-immunohistochemical study of RANKL, RANK, OPG: an experimental study in rats. Lasers Surg Med. 2007 Jun;39(5):441-50. doi: 10.1002/lsm.20508. PMID 17523169
- [Background] Amid R, Kadkhodazadeh M, Ahsaie MG, Hakakzadeh A. Effect of low level laser therapy on proliferation and differentiation of the cells contributing in bone regeneration. J Lasers Med Sci. 2014 Fall;5(4):163-70. PMID 25653816
- [Derived] Bozkaya S, Uraz A, Guler B, Kahraman SA, Turhan Bal B. The stability of implants and microbiological effects following photobiomodulation therapy with one-stage placement: A randomized, controlled, single-blinded, and split-mouth clinical study. Clin Implant Dent Relat Res. 2021 Jun;23(3):329-340. doi: 10.1111/cid.12999. Epub 2021 Apr 14. PMID 33851765